CLINICAL TRIAL: NCT01548365
Title: Impact of an Infusion Therapy Nursing Expert Service on Length of Stay, Clinical Results of Venous Access Devices and Satisfaction on Patients With Long Intravenous Therapy Prescription.
Brief Title: Impact of an Infusion Therapy Nursing Expert Service on Length of Stay and Clinical Results of Venous Access Devices
Acronym: ETI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Basque Health Service (Other Government)
Collaborators: KRONIKGUNE Cronicity Research Centre (Unknown)
Responsible Party: Principal Investigator, Lucia Garate Echenique, Nursing Research Supervisor, Basque Health Service
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: ITNE01
Record Dates: First submitted 2012-03-05; First posted 2012-03-08 (Estimated); Last update posted 2013-09-23 (Estimated); Status verified 2013-09

CONDITIONS: Patients With Prolonged Intravenous Therapy
Keywords: Nursing Services; Catheterization, Central Venous; Catheters Indwelling; Catheterization, Peripheral

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): routine care for the selection, placement and maintenance of venous access devices (VAD).
- Infusion Therapy Nursing Expert (Experimental): Patients in this group will receive the infusion therapy nursing expert (ITNE) service.
  Interventions: Other: Infusion therapy nursing expert service

INTERVENTIONS:
Other: Infusion therapy nursing expert service — The ITNE will assess the patient and treatment characteristics and use an evidence based decision making algorithm for the selection of the most suitable VAD.
  If the VAD needed is a PICC or a midline ITNE will place it following hospital's protocols. If needed, ITNE will also educate and support patients and next of keens in the maintenance of the device at home.
  If other devices such as peripheral catheters, central venous catheters (jugular or subclavian) or venous subcutaneous reservoirs are the preferable VADs for patients and treatment conditions, ITNE will work together with health professionals in charge of patients to activate the usual procedures to place the according device.
  Arms: Infusion Therapy Nursing Expert

SUMMARY:
The purpose of this study is to determine whether an infusion therapy nursing expert service is effective in decreasing hospital length of stay, improving the clinical results of venous access devices and increasing patient satisfaction with venous access.

ELIGIBILITY:
Inclusion Criteria:

* Require an estimated long prescription of intravenous treatment. These treatments may be of fluid therapy, pharmacological, nutritional or hemotherapy.

  * Estimation of 7 days or more of continuous intravenous therapy.
  * Estimation of an intermittent intravenous therapy of less than a week, but on a monthly basis or less and a total estimated duration superior to 3 months.
* Be patient at Araba University Hospital

Exclusion Criteria:

* To have a central venous catheter indwelled
* MRSA (Methicillin Resistant Staphylococcus Aureus)
* Younger than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2012-03; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Hospital Length of Stay | 3 months

SECONDARY OUTCOMES:
Venous Access Devices reaching end of treatment | 3 months
Incidence of complications derived from VAD | 3 months
Patients receiving intravenous therapy at home | 3 months
Patient satisfaction with VAD | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Lucia Garate, MsC, Principal Investigator — Basque Health Service
Locations (1):
- Araba University Hospital, Vitoria-Gasteiz, Araba, Spain